CLINICAL TRIAL: NCT02358967
Title: Palm Tocotrienols in Chronic Hemodialysis (PATCH Study)
Brief Title: Palm Tocotrienols in Chronic Hemodialysis (USA)
Acronym: PATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: DaVita, Inc. (Industry); Great Lakes Dialysis, LLC (Other); National University of Malaysia (Other); Universiti Putra Malaysia (Other); Ministry of Health, Malaysia (Other Government); National Kidney Foundation, United States (Other); PEMANDU (Unknown); Henry Ford Hospital (Other); Kidney Foundation Hospital and Research Institute, Bangladesh (Other); Fortis Hospital, India (Other)
Responsible Party: Principal Investigator, Pramod Khosla, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 123314MP4F
Record Dates: First submitted 2015-01-30; First posted 2015-02-09 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: End Stage Renal Disease; Chronic Kidney Disease
Keywords: ESRD; dyslipidemia; oxidative stress; inflammation; Hemodialysis; CKD
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Dyslipidemias; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Standard renal care + 300 mg placebo daily for 1 year
  Interventions: Dietary Supplement: Placebo
- Treatment (Active Comparator): Standard renal care + 300 mg TRF daily for 1 year
  Interventions: Dietary Supplement: TRF (Tocotrienol-rich-fraction)

INTERVENTIONS:
Dietary Supplement: TRF (Tocotrienol-rich-fraction) — 2 x 150 mg capsules
  Other Names: Tocotrienols are a naturally ocurring form of Vitamin E
  Arms: Treatment
Dietary Supplement: Placebo — 2 x 150 mg capsules
  Arms: Placebo

SUMMARY:
Patients undergoing chronic hemodialysis are at increased risk for cardiovascular disease, attributed in part to increased oxidative stress, inflammation and dyslipidemia. Intervention with a naturally occurring dietary supplement may improve certain biomarkers of inflammation and oxidative stress and improve the lipid profile.

DETAILED DESCRIPTION:
End stage renal disease (ESRD) patients who are undergoing hemodialysis (HD) have higher levels of blood markers which the body makes in response to increased stress and injury. An increase in these markers has been shown to be related to cardiovascular disease and death in ESRD patients. It is believed that taking antioxidants (e.g. Vitamin E) may decrease these markers. In a previous study in ESRD patients on HD, consumption of a Vitamin E tocotrienol-rich fraction (TRF) was found to improve some of these markers. The current study will follow a larger group of patients for a longer time period (1 year) and document effects on additional markers

The study will document the extent to which supplementation with TRF will improve markers of inflammation, oxidative stress as well as blood lipids in ESRD patients on chronic HD as compared to a placebo. Additionally, the study will aim to document any improvement in Restless Legs Syndrome - tingling sensation in the legs - (RLS) with TRF, based on a standard questionnaire.

The study will last for 15 months. At the start of the study basic patient information will be evaluated related to their monthly dialysis labs, inflammation and oxidative stress markers as well as general information about the patients in relation to their kidney disease. Patients will then be randomized into one of two groups. One group will receive TRF, daily, for 12 months while the second group will receive placebo, daily, for 12 months. Capsules will be administered in the dialysis clinic/unit at the start of each dialysis session (thrice weekly), while patients will be provided capsules to be consumed at home for the remaining four days of each week.

During the 12 month treatment period, patients will be questioned every three months at their dialysis units by study staff to obtain information on dialysis labs, medical condition, hospitalizations, and to check to see if they are taking the study capsules.

As part of their routine standard care, patients will continue to have monthly blood draws. For the purposes of this study, at each trimonthly blood draw, we will obtain additional blood to examine the markers related to oxidative stress, inflammation and lipids. A blood sample will also be collected at 15 months (3 months after patients stop taking capsules). Therefore over the course of the entire study, blood will obtained at baseline and 3, 6, 9 and 12 months (plus the 15 month follow-up sample).

At each trimonthly blood draw including the follow-up visit at 15 months, patients will also be verbally administered a Restless Legs Syndrome Questionnaire. In addition a dietitian member of the research team will administer a 24 hr diet recall questionnaire

Sample size was based on inflammatory markers (hsCRp and IL-6) as reported in earlier studies and a sample size of 175 per group was estimated to achieve a 80% power at p=0.05 significance level. Thus accounting for potential drop-outs over the 1 year of the study, target is recruitment of 400 patients total (200 for each group) in Detroit, MI.

(A similar study, following a similar protocol and using the same study design and intervention will recruit 400 patients total (200 for each group) in Kuala Lumpur, Malaysia).

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 years and above. Undergoing chronic hemodialysis treatment for more than 3 months (life expectancy > 1 year).
* Able and willing to comply with all trial requirements.
* Willing to allow his or her /Physician/Nephrologist/General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* History of functional kidney transplant 6 months before study entry; anticipated live donor kidney transplant over the study duration;
* Participants who are taking vitamin E- containing supplements >60 IU/d during the past 30 days
* History of poor adherence to hemodialysis or medical regimen
* Participants who are currently on active treatment for cancer, excluding basal cell carcinoma of the skin
* Participants who have been diagnosed as HIV/AIDS and/or on the anti-HIV therapy. (HIV seropositivity is not an exclusion criterion)
* Patients taking anti-inflammatory medication, except aspirin<325 mg/d, over the past 30 days
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Participants who are receiving nutritional support (i.e. enteral and intra-venous route)
* Patients using a temporary catheter for dialysis access at baseline or patients receiving a graft/fistula within the 6-month study period
* More than two hospitalizations within the last 90 days or one hospitalization within the 30 days preceding enrollment
* Any other significant disease or disorder which, in the opinion of their nephrologist, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | Every 3 months, upto 15 months
  measurement of hsCRP from blood samples

SECONDARY OUTCOMES:
Plasma lipids | Every 3 months, upto 15 months
  TC, TAG, HDL-C (all in mg/dL plasma)
Restless Legs Syndrome | Every 3 months, upto 15 months
  A questionnaire (Restless Legs Syndrome Rating Scale). The RLS questionnaire consists of 10 questions, each can be scored from 0 to 4 points. The final score can range from 0 to 40 points.
Dietary history | Every 3 months, upto 15 months
  A diet questionnaire based on a 24 h diet recall

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Khosla, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Background] Daud ZA, Tubie B, Sheyman M, Osia R, Adams J, Tubie S, Khosla P. Vitamin E tocotrienol supplementation improves lipid profiles in chronic hemodialysis patients. Vasc Health Risk Manag. 2013;9:747-61. doi: 10.2147/VHRM.S51710. Epub 2013 Nov 28. PMID 24348043
- [Background] Daud ZA, Tubie B, Adams J, Quainton T, Osia R, Tubie S, Kaur D, Khosla P, Sheyman M. Effects of protein and omega-3 supplementation, provided during regular dialysis sessions, on nutritional and inflammatory indices in hemodialysis patients. Vasc Health Risk Manag. 2012;8:187-95. doi: 10.2147/VHRM.S28739. Epub 2012 Mar 20. PMID 22536073